CLINICAL TRIAL: NCT05660018
Title: TMS Related Biomarker Assessments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Xiaoming Du, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: HP-00103592
Record Dates: First submitted 2022-12-02; First posted 2022-12-21 (Actual); Results first posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia Schizoaffective; Schizophrenia
Keywords: schizophrenia; Transcranial magnetic stimulation
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active rTMS first and sham rTMS second (Other): Participants in this arm will receive active rTMS in one visit first, then receive sham rTMS in another visit.
  Interventions: Device: active rTMS first, then sham rTMS
- Sham rTMS first and active rTMS second (Other): Participants in this arm will receive sham rTMS in one visit first, then receive active rTMS in another visit.
  Interventions: Device: sham rTMS first, then active rTMS

INTERVENTIONS:
Device: active rTMS first, then sham rTMS — Active rTMS is delivered on the first visit, then sham rTMS is delivered on the second visit.
  Arms: Active rTMS first and sham rTMS second
Device: sham rTMS first, then active rTMS — Sham rTMS is delivered on the first visit, then active rTMS is delivered on the second visit.
  Arms: Sham rTMS first and active rTMS second

SUMMARY:
Patients with schizophrenia spectrum disorder (SSD) will be exposed to active and sham repetitive transcranial magnetic stimulation (rTMS) in separate sessions. SSD-related biomarkers will be assessed before and after the rTMS administration.

DETAILED DESCRIPTION:
Electrical neural oscillations of the brain can be measured at many levels, ranging from single cell to local field potentials in animals, to large-scale synchronized activities in the human scalp. New evidence suggests that there may be common underlying abnormalities in oscillatory activities that are associated with schizophrenia-related cognitive and functional impairments. There is currently no treatment for these electrical oscillation dysfunctions. Transcranial magnetic stimulation (TMS) provides a non-invasive means for altering brain electrical neural activity. TMS has been approved by FDA for the treatment of depression and many other mental disorders. It has been used in a wide range of clinical research, especially in neurology and psychiatry. The investigators aim to develop TMS paradigms that will modulate brain responses during basic sensory to more complex cognitive performance and determine the parameters in anatomic locations and TMS modalities that may effectively and safely modulate neural activities. If the current experiments successfully identified TMS methods/paradigms that improve neural oscillation and cognitive performances in schizophrenia patients, in the future (not part of the current protocol), the investigators can then develop specific TMS treatment that may correct abnormal brain function and improve cognition and clinical symptoms of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female between ages 18-65
* Ability to give written informed consent (age 18 or above)
* Diagnosed with schizophrenia-spectrum disorder and Evaluation to Sign Consent (ESC) above10.

Exclusion Criteria:

* Any history of seizures.
* Significant alcohol or other drug use (substance dependence within 6 months or substance abuse within 1 month) other than nicotine or marijuana dependence.
* Any major medical illnesses that may affect normal brain functioning. Examples of these conditions include, but not limited to, stroke, CNS infection or tumor, other significant brain neurological conditions.
* Taking > 400 mg clozapine/day
* Failed TMS screening questionnaire
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed.
* History of head injury with loss of consciousness over 10 minutes; history of brain surgery
* Can not refrain from using alcohol and/or marijuana 24 hours or more & cigarette smoking half and hour or more prior to experiments.
* Woman who is pregnant (child-bearing potential but not on contraceptive and missing menstrual period; or by self report; or by positive pregnancy test) or has had unprotected sexual intercourse without birth control in the last 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Du, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active rTMS First and Sham rTMS Second | Sham rTMS First and Active rTMS Second
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active rTMS First and Sham rTMS Second | Sham rTMS First and Active rTMS Second | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (18.2) | 39.2 (16.2) | 39.0 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change of Resting-state Functional Connectivity (rsFC) by Active and Sham rTMS
Description: The strength of rsFC was first defined by correlation coefficient (r). Because the distribution of r values is highly skewed, z scores (normally distributed) were computed via fisher r-to-z transform. The z score central value (i.e., z score of 0) represents no relationship between the two brain regions. A positive (negative) z score indicates a positive (negative) association between the two brain regions. Stronger rsFC (i.e., larger positive z score) was related to stronger connection between the two brain regions. The differences of rsFC between active and sham were reported. A positive (negative) value of rsFC change suggests the rsFC was enhanced (weakened) by active TMS.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: z score of functional connectivity
Groups:
- Active rTMS: Participants who received active rTMS in either the first or the second visit.
- Sham rTMS: Participants who received sham rTMS in either the first or second visit.
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
z score of functional connectivity | 0.018 (0.018) | 0.007 (0.027)

2. Primary Outcome: Change of Mismatch Negativity (MMN) From Electroencephalography (EEG) Signals by Active and Sham rTMS
Description: TMS effect is explored by comparing MMN changes from active and sham rTMS. MMN is measured by subtracting the averaged EEG response to a set of standard stimuli from the averaged response to rarer deviant stimuli, and taking the amplitude of this difference wave in a given time window. The differences of MMN between active and sham were reported. A negative (positive) value of rsFC change suggests the MMN was enhanced (weakened) by active TMS.
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: microvolts
Groups:
- Sham rTMS: Participants who received sham rTMS in either the first or the second visit.
Arm/Group | Active rTMS | Sham rTMS
Number analyzed (Participants) | 10 | 10
microvolts | -0.106 (0.367) | 0.044 (0.217)

ADVERSE EVENTS:
Time Frame: From baseline to the time when the participant completes or quits the study (up to 1 month).
Arm/Group | Active rTMS | Sham rTMS
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/18/NCT05660018/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT05660018/ICF_002.pdf